CLINICAL TRIAL: NCT04697069
Title: A Phase 2a, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of ANB019 in the Treatment of Acneiform Rash in Subjects With Neoplasm Receiving EGFRi or MEKi Therapy
Brief Title: A Study to Evaluate of the Efficacy and Safety of Imsidolimab (ANB019) in the Treatment of Acneiform Rash
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Administrative Reason
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANB019-207; 2020-003494-22 (EudraCT Number)
Record Dates: First submitted 2020-12-23; First posted 2021-01-06 (Actual); Results first posted 2023-01-09 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2022-12

CONDITIONS: Acneiform Eruptions
Keywords: IL-36 receptor; Interleukin 36; Imsidolimab
MeSH Terms: conditions — Acneiform Eruptions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ANB019 (Experimental): Participants received a starting dose of 400 milligrams (mg) of imsidolimab on Day 1 followed by 200 mg imsidolimab every 4 weeks (Days 29, 57 and 85) by subcutaneous injection.
  Interventions: Biological: Imsidolimab
- Placebo (Placebo Comparator): Participants received imsidolimab matching placebo on Day 1 and thereafter, every 4 weeks (Days 29, 57 and 85) by subcutaneous injection.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Imsidolimab — Humanized monoclonal antibody
  Other Names: ANB019
  Arms: ANB019
Biological: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Efficacy and Safety of imsidolimab in participants with epidermal growth factor receptor inhibitor (EGFRi)/mitogen-activated protein (MAP)/extracellular signal-regulated kinase (ERK) kinase inhibitor (MEKi)-associated acneiform Rash

DETAILED DESCRIPTION:
This study is a Phase 2a, multicenter, randomized, double-blind, placebo-controlled study to evaluate the efficacy, safety, and tolerability of imsidolimab compared with placebo in cancer participants with EGFRi/MEKi-associated acneiform rash. This study will also characterize the pharmacokinetic (PK) profile of imsidolimab and explore the immune response to imsidolimab in participants with EGFRi/MEKi-associated acneiform rash.

ELIGIBILITY:
Inclusion Criteria:

* Participant has cancer
* Participant is treated with an oral or injectable Food and Drug Administration (FDA)-approved EGFRi or MEKi therapy
* Participant has EGFRi/MEKi-related acneiform rash of Grade ≥ 2 as per common terminology criteria for adverse events (CTCAE) version 5.0, and ≥ 20 inflammatory lesions on the face at screening and Day 1.

Exclusion Criteria:

* Participant has infected EGFRi/MEKi-associated acneiform rash according to investigator's evaluation.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-05-04 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2021-12-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (18):
- United States (5):
  - Site 102, Tampa, Florida
  - Site 106, Boston, Massachusetts
  - Site 101, St Louis, Missouri
  - Site 105, Columbus, Ohio
  - Site 103, Houston, Texas
- Czechia (4):
  - Site 302, New Town, Praha 2
  - Site 303, Brno
  - Site 301, Olomouc
  - Site 304, Plzen-Bory
- Georgia (5):
  - Site 404, Batumi
  - Site 402, Tbilisi
  - Site 403, Tbilisi
  - Site 405, Tbilisi
  - Site 401, Tbilisi
- Site 601, Riga, Latvia
- Poland (3):
  - Site 204, Gliwice
  - Site 203, Poznan
  - Site 201, Szczecin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with neoplasms who were receiving epidermal growth factor inhibitors or mitogen-activated protein/extracellular signal regulated kinase inhibitor were enrolled into the study.
Pre-assignment Details: 11 participants were screened for eligibility and 4 participants were randomized into the study.
Groups:
- Imsidolimab: Participants received a starting dose of 400 milligrams (mg) of imsidolimab on Day 1 followed by 200 mg imsidolimab every 4 weeks (Days 29, 57 and 85) by subcutaneous injection.
Period: Overall Study
Arm/Group | Imsidolimab | Placebo
Started | 2 | 2
Completed | 0 | 0
Not Completed | 2 | 2
Not completed — Withdrew consent due to possible/perceived lack of efficacy by participants | 0 | 1
Not completed — Study termination | 2 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) analysis set included all randomized participants.
Groups:
- Imsidolimab: Participants received a starting dose of 400 mg of imsidolimab on Day 1 followed by 200 mg imsidolimab every 4 weeks (Days 29, 57 and 85) by subcutaneous injection.
- Total: Total of all reporting groups
Arm/Group | Imsidolimab | Placebo | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.0 (9.90) | 65.0 (2.83) | 57.5 (10.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Facial Inflammatory Lesion Count (Papules and Pustules) at Week 8
Description: The number of facial inflammatory lesions (papules and pustules) on the face (excluding the neck and scalp area) was counted. Papule was a small, solid elevation 5 millimeters (mm) or less in diameter. Pastule was a small, circumscribed elevation of the skin that contains yellow-white exudate.
Time Frame: Baseline, Week 8
Population: Due to early study termination, no participant was evaluated in the imsidolimab group and 1 participant was evaluated in the placebo group. Since only 1 participant was evaluated, results were not reported for the protection of personal data and to avoid re-identification.
Arm/Group | Imsidolimab | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Percent Change From Baseline in Facial Inflammatory Lesion Count (Papules and Pustules) at Week 8
Description: The number of facial inflammatory lesions (papules and pustules) on the face (excluding the neck and scalp area) was counted. Papule was a small, solid elevation 5 mm or less in diameter. Pastule was a small, circumscribed elevation of the skin that contains yellow-white exudate.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Arm/Group | Imsidolimab | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Percentage of Participants With an Improvement of at Least 1 Grade From Baseline in Acneiform Rash Common Terminology Criteria for Adverse Events (CTCAE) Grading Scale at Week 8
Description: The acneiform rash CTCAE grading scale of severity was 6-point scale ranging from 0-5.
  Scale 0=no evidence of rash. Scale 1= papules and/or pustules covering <10% body surface area (BSA), which may or may not be associated with symptoms of pruritus or tenderness.
  Scale 2=papules and/or pustules covering 10-30% BSA, which may or may not be associated with symptoms of pruritus or tenderness; associated with psychosocial impact; limiting instrumental activities of daily living (ADL); papules and/or pustules covering >30% BSA with or without mild symptoms.
  Scale 3=papules and/or pustules covering >30% BSA with moderate or severe symptoms; limiting self-care ADL; associated with local superinfection with oral antibiotics.
  Scale 4=life-threatening consequences; papules and/or pustules covering any %BSA, which may or may not be associated with symptoms of pruritus or tenderness and are associated with extensive superinfection with intravenous (IV) antibiotics indicated.
  Scale 5=death.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Arm/Group | Imsidolimab | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Time to First Response of 1 Grade Improvement From Baseline on the Acneiform Rash CTCAE Grading Scale
Description: Time to first response of 1 grade improvement from baseline on the acneiform rash CTCAE grading scale: Date of the first response of 1 grade improvement from baseline on the acneiform rash CTCAE grading scale - Date of the first dose of study treatment (or from randomization for any participant randomized but not treated) + 1.
Time Frame: Baseline up to 55 days
Population: as for outcome 1
Arm/Group | Imsidolimab | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Percentage of Participants With an Improvement of at Least 1 Grade From Baseline in Acneiform Rash Modified Multinational Association for Supportive Care in Cancer (MASCC) EGFRi Skin Toxicity Tool (MESTT) Grading Scale (Total Score) at Week 8
Description: The MESTT grading scale of the acneiform rash severity was a 3-point scale ranging from 1 to 3:
  Scale 1 = 1A: papules or pustules ≤5; OR 1 area of erythema or edema <1 centimeter (cm) in size. 1B: papules or pustules ≤5; OR 1 area of erythema or edema <1 cm in size; AND pain or pruritus.
  Scale 2 = 2A: papules or pustules 6-20; OR 2-5 areas of erythema or edema <1 cm in size. 2B: Papules or pustules 6-20; OR 2-5 areas of erythema or edema <1 cm in size; AND pain, pruritus, or effect on emotions or functioning.
  Scale 3 = 3A: papules or pustules > 20; OR more than 5 areas of erythema or edema <1 cm in size. 3B: papules or pustules > 20; OR more than 5 areas of erythema or edema <1 cm in size; AND pain, pruritus, or effect on emotions or functioning.
  Grading was performed individually for the face, scalp, chest, and back. The sum of all body region scores yielded the total score (range: 4 to 12).
Time Frame: Baseline, Week 8
Population: as for outcome 1
Arm/Group | Imsidolimab | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Time to First Response of 1 Grade Improvement From Baseline on the Acneiform Rash Modified MESTT Grading Scale (Total Score)
Description: Time to first response of 1 grade improvement from baseline on the acneiform rash modified MESTT grading scale (total score): Date of onset of the first response of 1 grade improvement from baseline on the acneiform rash modified MESTT grading scale (total score) - Date of the first dose of study treatment (or from randomization for any participant randomized but not treated) + 1.
Time Frame: Baseline to 55 days
Population: as for outcome 1
Arm/Group | Imsidolimab | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Percentage of Participants With an Improvement of at Least 1 Grade From Baseline in Acneiform Rash Modified MESTT Grading Scale (Facial Assessment) at Week 8
Description: The MESTT grading scale of the acneiform rash severity was a 3-point scale ranging from 1 to 3:
  Scale 1 = 1A: papules or pustules ≤5; OR 1 area of erythema or edema <1cm in size. 1B: papules or pustules ≤5; OR 1 area of erythema or edema <1 cm in size; AND pain or pruritus.
  Scale 2 = 2A: papules or pustules 6-20; OR 2-5 areas of erythema or edema <1 cm in size. 2B: Papules or pustules 6-20; OR 2-5 areas of erythema or edema <1 cm in size; AND pain, pruritus, or effect on emotions or functioning.
  Scale 3 = 3A: papules or pustules > 20; OR more than 5 areas of erythema or edema <1 cm in size. 3B: papules or pustules > 20; OR more than 5 areas of erythema or edema <1 cm in size; AND pain, pruritus, or effect on emotions or functioning.
  Grading was performed individually for the face. The score ranged from 1 to 3.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Arm/Group | Imsidolimab | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Time to First Response of 1 Grade Improvement From Baseline on the Acneiform Rash Modified MESTT Grading Scale (Facial Assessment)
Description: Time to first response of 1 grade improvement from baseline on the acneiform rash modified MESTT grading scale (facial assessment): Date of onset of the first response of 1 grade improvement from baseline on the acneiform rash modified MESTT grading scale (facial assessment) - Date of the first dose of study treatment (or from randomization for any participant randomized but not treated) + 1.
Time Frame: Baseline to 55 days
Population: as for outcome 1
Arm/Group | Imsidolimab | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change From Baseline in Pruritus Numeric Rating Scale (NRS) at Week 8
Description: The intensity of pruritus was evaluated by asking participants to assign a numerical score representing the worst intensity over the last 24 hours of their symptoms on a scale from 0 to 10, with 0 indicating no itch and 10 indicating the worst imaginable itch.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Arm/Group | Imsidolimab | Placebo
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Percent Change From Baseline in Pruritus NRS at Week 8
Description: as for outcome 9
Time Frame: Baseline, Week 8
Population: as for outcome 1
Arm/Group | Imsidolimab | Placebo
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Change From Baseline in Pain NRS at Week 8
Description: The intensity of pain was evaluated by asking participants to assign a numerical score representing the worst intensity over the last 24 hours of their symptoms on a scale from 0 to 10, with 0 indicating no pain and 10 indicating the worst imaginable pain.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Arm/Group | Imsidolimab | Placebo
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Percent Change From Baseline in Pain NRS at Week 8
Description: as for outcome 11
Time Frame: Baseline, Week 8
Population: as for outcome 1
Arm/Group | Imsidolimab | Placebo
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy - Epidermal Growth Factor Receptor Inhibitor 18 (FACT-EGFRi-18) at Week 8
Description: The FACT-EGFRi-18 was an 18-item likert-scaled questionnaire, arranged in three dimensions: physical (seven items), social/emotional (six items), and functional well-being (five items). The response scores ranged from 0 (not at all) to 4 (very much).
  The total score was obtained by multiplying the sum of the subscale by the number of items in the scale (18), and then dividing by the number of items actually answered.
  The total score ranged from 0-72 with a higher score represented a high level of symptomatology (problems).
Time Frame: Baseline, Week 8
Population: as for outcome 1
Arm/Group | Imsidolimab | Placebo
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events
Description: An adverse event (AE) was any untoward medical occurrence in a participant temporally associated with the use of a study treatment, whether or not considered related to study treatment. An AE could therefore be any unfavorable and unintended sign (including abnormal laboratory finding), symptom, or disease temporally associated with use of study treatment that did not necessarily have a causal relationship with this treatment. An AE was considered "serious" if there was any of the following outcomes: death, life-threatening, Inpatient hospitalization or prolongation of existing hospitalization, persistent or significant incapacity or substantial disruption of ability to conduct normal life functions, congenital anomaly/birth defect, other important medical events. An AE was considered treatment-emergent if the date of onset was during or after first dose of study treatment, or if the AE present at baseline worsened in either intensity or frequency after first dose of study treatment.
Time Frame: From first dose to 55 days
Population: Safety analysis set included all randomized participants who received at least 1 dose of imsidolimab or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Imsidolimab | Placebo
Number analyzed (Participants) | 2 | 2
Participants
  Any TEAEs | 0 | 2
  Serious TEAEs | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose to 55 days
Description: Safety analysis set included all randomized participants who received at least 1 dose of imsidolimab or placebo.
Arm/Group | Imsidolimab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Imsidolimab (N=2) | Placebo (N=2)
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Electrocardiogram T wave inversion (Investigations) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-08-05): https://cdn.clinicaltrials.gov/large-docs/69/NCT04697069/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-11): https://cdn.clinicaltrials.gov/large-docs/69/NCT04697069/SAP_001.pdf